CLINICAL TRIAL: NCT05980871
Title: Treatment Responses of Early Syphilis to Single-dose Ceftriaxone Plus Doxycycline Versus Single-dose Benzathine Penicillin G Plus Doxycycline in PLWH
Brief Title: Treatment Responses of Early Syphilis to Ceftriaxone Plus Doxycycline
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202206138MIND
Record Dates: First submitted 2023-03-08; First posted 2023-08-08 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Early Syphilis
MeSH Terms: conditions — Syphilis | interventions — Doxycycline; Ceftriaxone; Penicillin G

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- single-dose ceftriaxone plus doxycycline (Active Comparator): single-dose ceftriaxone (1g intramuscularly once) plus doxycycline (100 mg orally twice daily for 7 days)
  Interventions: Drug: Doxycycline; Drug: Ceftriaxone
- single-dose BPG plus doxycycline (Active Comparator): single-dose BPG (2.4 MU intramuscularly once) plus doxycycline (100 mg orally twice daily for 7 days)
  Interventions: Drug: Doxycycline; Drug: benzathine penicillin G

INTERVENTIONS:
Drug: Doxycycline — doxycycline (100 mg orally twice daily for 7 days)
Drug: Ceftriaxone — Ceftriaxone (1g intramuscularly once)
  Arms: single-dose ceftriaxone plus doxycycline
Drug: benzathine penicillin G — benzathine penicillin G (2.4 MU intramuscularly once)
  Arms: single-dose BPG plus doxycycline

SUMMARY:
In a prospective study investigating the prevalence of STIs among at-risk PLWH, the prevalence of Chlamydia trachomatis and N. gonorrhoeae was 24.7% and 12.1%, respectively. Surprisingly, the study found high rates of C. trachomatis and/or N. gonorrhoeae co-infections in PLWH with recent hepatitis C virus (HCV) infection (50%), HBsAg positivity (44%), and early syphilis (36%). Considering the high rate of sexually transmitted co-infections, combination therapy of single-dose ceftriaxone plus 7-day doxycycline for early syphilis may provide convenience and benefit to treatment of N. gonorrhoeae and C. trachomatis co-infections at a single clinic encounter. In the present study, this study aim to compare the efficacy of ceftriaxone plus doxycycline versus BPG plus doxycycline as the treatment for early syphilis among PLWH.

DETAILED DESCRIPTION:
Enrolled criteria:

1. PLWH aged 20 years or more
2. PLWH with early syphilis (i.e. primary, secondary, or early latent syphilis), confirmed by a positive rapid plasma reagin (RPR) titer with a reactive Treponema pallidum particle agglutination (TPPA) assay.
3. PLWH has provided informed consent *A participant with repeated syphilis can be repeated enrolled after signing an informed consent if the previous episode of early syphilis was successfully treated with achieving at least a 4-fold decrease in RPR titers and 48-week follow-up is completed.

Exclusion criteria:

1. PLWH with RPR titers of less than 4
2. Exposure to antibiotics with activity against T. pallidum, such as penicillins, third-generation cephems, doxycycline, or macrolides, within the preceding 4 weeks
3. A known or suspected infection other than syphilis requiring additional treatment with an antimicrobial active against T. pallidum
4. A history of intolerance to penicillin, ceftriaxone, or doxycycline
5. Pregnancy

Primary outcome:

Serologic response at month 6 (defined as either a 4-fold or greater decline in RPR titer compared to baseline or being RPR-nonreactive)

Secondary outcomes:

1. Microbiologic response of syphilis (defined as T. pallidum PCR Ct value >38) at week 4
2. Microbiologic response of bacterial STIs (defined as negative PCR results) at week 4
3. Serologic response at months 3 and 12
4. Safety of study treatment recorded by using a diary (all adverse events will be coded and graded according to Common Terminology Criteria for Adverse Events [CTCAE] v4.0.)
5. Adherence evaluation (the noting of tablet intake in the diary for the 7 days of the treatment period)

ELIGIBILITY:
Inclusion Criteria:

* PLWH aged 20 years or more
* PLWH with early syphilis (i.e. primary, secondary, or early latent syphilis), confirmed by a positive rapid plasma reagin (RPR) titer with a reactive Treponema pallidum particle agglutination (TPPA) assay.
* PLWH has provided informed consent

Exclusion Criteria:

* PLWH with RPR titers of less than 4
* Exposure to antibiotics with activity against T. pallidum, such as penicillins, third- generation cephems, doxycycline, or macrolides, within the preceding 4 weeks
* A known or suspected infection other than syphilis requiring additional treatment with an antimicrobial active against T. pallidum
* A history of intolerance to penicillin, ceftriaxone, or doxycycline
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Rate of serologic response at month 6 | Month 6
  Serologic response is defined as either a 4-fold or greater decline in RPR titer compared to baseline or being RPR-nonreactive

SECONDARY OUTCOMES:
Rate of microbiologic response of syphilis at week 4 | Week 4
  Microbiologic response of syphilis is defined as T. pallidum PCR Ct value >38
Rate of microbiologic response of bacterial STIs at week 4 | Week 4
  Microbiologic response of bacterial STIs is defined as negative PCR results
Rate of serologic response at months 3 and 12 | Months 3 and 12
  Serologic response is defined as either a 4-fold or greater decline in RPR titer compared to baseline or being RPR-nonreactive

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Yin Lin, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Kuan-Yin Lin, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No